CLINICAL TRIAL: NCT00964184
Title: Phenotypic and Genetic Correlates of Diabetes (Non-Type 1) in Young Non-Obese Asian Indians in North India and A Study to Evaluate the Efficacy of Sitagliptin (DPP-4 Inhibitor) in a Sub-group of the Study Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Responsible Party: Principal Investigator, Dr Anoop Misra, Director, Diabetes, Obesity and Metabolic Disorders, Diabetes Foundation, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LeanDM-01
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Maturity onset diabetes of the young 3 protein, human
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Maturity-Onset Diabetes of the Young, Type 3 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug (Experimental): 1 gm metformin per day
  Interventions: Drug: Metformin
- control (Other): lifestyle intervention
  Interventions: Behavioral: Lifestyle modification

INTERVENTIONS:
Drug: Metformin
  Arms: Drug
Behavioral: Lifestyle modification
  Arms: control

SUMMARY:
This is a phase IV study of 3.5 years duration to evaluate the phenotypic and genetic correlates of diabetes (non-Type 1 in young non-obese Asian Indians in North India and pilot case control study to evaluate the efficacy of sitagliptin (DPP-4 inhibitor) in a sub-group of the study population.

DETAILED DESCRIPTION:
A phase IV on T2DM with BMI < 25 kg/m2 and age 14-40 years.

Primary Objectives:

* To investigate phenotype (body composition, anthropometry, pancreatic imaging and endocrine function, insulin resistance, autoantibodies, and other biochemical variables) and genetic (known mutations and polymorphisms) correlates in young (age 14-40 years) diabetic patients (non-type 1).

Secondary Objectives:

* To study anthropometric and body fat distribution including truncal fat, subcutaneous and intra-abdominal fat in non-obese young patients with diabetes (non-type 1).
* To study whether insulin secretion, insulin resistance or a combination of both is/are the predominant defect(s) in non-obese young diabetics (non-type 1).
* To study the prevalence of autoimmunity and/or specific genetic abnormalities in this subgroup of diabetics.
* To estimate approximate prevalence of diagnostic subcategories based on the sample of population, and profile of complications in each category.
* To propose rational use of specialized investigations (e.g. GAD65, HNF-1α mutations etc) while investigating a newly diagnosed young diabetic.
* To determine the rational therapeutic option and prognosis in this sub-population of diabetics based on anthropometric, biochemical, and etiological profiles.
* Sample size: 205 patients to be enrolled and 120 patients to be enrolled for sub group study

ELIGIBILITY:
Inclusion Criteria:

* Young (18 to 40 years) patients with diabetes (not on insulin therapy) during the past 6 months and having BMI <25 kg/m2.
* Drug naïve patients
* Patients on mono-therapy with metformin (< 1g/day).

Exclusion Criteria:

* Type 1 diabetes
* Type 2 Diabetes on any other oral hypoglycemic agent other than metformin
* Pregnancy or lactation
* Insulin or Sulfonylurea treatment within the past 3 months
* Has received any investigational drug with the past 60 days
* History of prior allergy or hypersensitivity to any drug (unless approved by investigator)
* HbA1c < 7.5% or > 8.5%.
* Unstable glycemic control, requiring addition of 2nd oral agent/insulin or frequent up-titration of dose of metformin.
* Any patient on insulin.
* Females of child bearing potential who are not using adequate contraception during the study period.
* Insulin dependent or history of ketoacidosis requiring hospitalization
* Acute infections
* Advanced end-organ damage (CLD, CRF etc.)
* Diabetes with clinically significant or advanced end-organ damage

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 133 (Actual)
Dates: Start 2009-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
HbA1c | 18 weeks
HbA1C | 12 weeks

SECONDARY OUTCOMES:
Assessment of safety profile of sitagliptin | 18 weeks
insulin | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Misra, Principal Investigator — Diabetes Foundation, India
Locations (1):
- Fortis Flt Lt Rajan Dhall Hospital, New Delhi, National Capital Territory of Delhi, India